CLINICAL TRIAL: NCT03168451
Title: American Indians STOp Smoking by Mobile Phone
Acronym: AI STOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Optum, Inc. (Industry)
Responsible Party: Principal Investigator, Dedra Buchwald, Director and Professor, Washington State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P20MD006871 (NIH)
Record Dates: First submitted 2017-01-30; First posted 2017-05-30 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-09

CONDITIONS: Tobacco Use Cessation
Keywords: text messaging
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Intervention Model Description: The intervention group will receive data collection messages and culturally tailored messages encouraging them to quit smoking. The control group will only receive data collection messages.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Members of the intervention group will receive culturally tailored text messages encouraging them to quit smoking. They will receive data collection text messages at 6, 12, 18, and 26 weeks post target quit date, assessing their current tobacco smoking behavior.
  Interventions: Behavioral: Culturally Tailored Text Messages
- Control (No Intervention): Members of the control group will receive data collection text messages at 6, 12, 18, and 26 weeks post target quit date, assessing their current tobacco smoking behavior.

INTERVENTIONS:
Behavioral: Culturally Tailored Text Messages — Members of the intervention group receive culturally tailored messages on the following schedule: 4 messages per day for 1 week prior to target quit date, 4 messages per day for 4 weeks following target quit date, 3 messages per week for 20 weeks following weeks.
  Arms: Intervention

SUMMARY:
In an attempt to reduce smoking-related health disparities, investigators will implement a text messaging-based smoking cessation intervention in collaboration with state quit lines. The approach is based on the successful STOMP (STOp smoking by Mobile Phone) program, a text messaging-based smoking cessation intervention among young Maori adults in New Zealand. Investigators will adapt the STOMP intervention, which will result in a new intervention known as AI STOMP (American Indians STOp smoking by Mobile Phone).The primary aim of the study is to determine the effectiveness of the AI-STOMP intervention in smoking cessation among American Indians.

DETAILED DESCRIPTION:
This is a randomized, single-blinded, controlled trial examining the effectiveness of a text messaging-based smoking cessation program among American Indian (AI) smokers who call state quit lines, in states with high AI populations. Participants will be randomized to either receive culturally-tailored text-messages to support smoking cessation or quit line's treatment as usual.

Participants will be recruited by Optum, the company who runs many state quit lines in the US. If - after answering some demographic questions for Optum from the following states: Alaska, Oklahoma, Wisconsin, Minnesota, and New Mexico - a person is found to be a AI/AN and 18+ years old, that person will be asked if they would like to receive information about the study. If they answer yes the WSU research team will receive their contact information from Optum via a secure email, and WSU researchers will send a text explaining the study in more detail and a link to the e-consent form.

Participants will also fill out 4 baseline questionnaires. After filling out baseline questionnaires, participants will be randomized to either the intervention group or the control group. Participants will be stratified into the intervention and control groups based on their age, gender, and Fagerstrom nicotine dependence score. Random permuted blocks will be used by on-campus research staff to manually assign participants to the two research groups.

All participants will begin receiving text messages one week before their chosen quit date.

ELIGIBILITY:
Inclusion Criteria:

* Identify as American Indian
* Be age 18 years or older
* Possess or have access to a mobile phone with text messaging capacity
* Be a current daily smoker; and
* Be interested in quitting smoking within the next 30 days

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 346 (Actual)
Dates: Start 2015-11-30 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who change smoking status as measured by self-report | 6, 12, 18, and 26 weeks after target quit date
  Number of participants who quit smoking while receiving text messages, as measured by self-report at 4 time points over 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dedra Buchwald, MD, Principal Investigator — Washington State University; Sterling McPherson, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University Coordinating Center, Spokane, Washington, United States

IPD SHARING:
Plan to Share IPD: No